CLINICAL TRIAL: NCT01566643
Title: Rabeprazole Based Sequential-Concommitant Hybrid Therapies for H. Pylori Infections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Collaborators: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Ming-Cheh Chen, Principal Investigator, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCRD100-16; IRB099-71 (Other: IRB of Buddhist Tzu Chi General Hospital)
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; antibiotic resistance; sequential-concomitant hybrid therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hybrid-10 (Experimental): RA3-RACM7: rabeprazole + amoxicillin x 3 days, then rabeprazole + amoxicillin + clarithromycin + metronidazole x 7 days.
  Interventions: Drug: RA3-RACM7
- Hybrid-12 (Experimental): RA5-RACM7: rabeprazole + amoxicillin x 5 days, then rabeprazole + amoxicillin + clarithromycin + metronidazole x 7 days
  Interventions: Drug: RA5-RACM7
- Hybrid-14 (Experimental): RA7-RACM7: rabeprazole + amoxicillin x 7 days, then rabeprazole + amoxicillin + clarithromycin + metronidazole x 7 days
  Interventions: Drug: RA7-RACM7

INTERVENTIONS:
Drug: RA5-RACM7 — rabeprazole 20mg bid + amoxicillin 1g bid treated for 5 days, then rabeprazole 20mg bid + amoxicillin 1g bid + clarithromycin 0.5g bid + metronidazole 0.5g bid for other 7 days
  Other Names: Pariet x 12 days.; Hiconcil x 12 days.; Klarid x 7 days.; Flagyl x 7 days.
  Arms: Hybrid-12
Drug: RA3-RACM7 — rabeprazole 20mg bid + amoxicillin 1g bid treated for 3 days, then rabeprazole 20mg bid + amoxicillin 1g bid + clarithromycin 0.5g bid + metronidazole 0.5g bid for other 7 days
  Other Names: Pariet x 10 days.; Hiconcil x 10 days.; Klarid x 7 days.; Flagyl x 7 days.
  Arms: Hybrid-10
Drug: RA7-RACM7 — rabeprazole 20mg bid + amoxicillin 1g bid treated for 7 days, then rabeprazole 20mg bid + amoxicillin 1g bid + clarithromycin 0.5g bid + metronidazole 0.5g bid for other 7 days
  Other Names: Pariet x 14 days.; Hiconcil x 14 days.; Klarid x 7 days.; Flagyl x 7 days.
  Arms: Hybrid-14

SUMMARY:
This prospective controlled randomized open-label clinical trial is designed to determine the optimal eradication rate of rabeprazole based sequential-concommitant hybrid therapies for adults infected with Helicobacter pylori in Eastern Taiwan. Enrolled patients will receive 3, 5 or 7 days of pre-concommitant (sequential part) treatment with rabeprazole + amoxicillin, then 7 days of concommitant treatment with rabeprazole + amoxicillin + clarithromycin + metronidazole.

DETAILED DESCRIPTION:
Background: Antimicrobial resistance has decreased the worldwide eradication rates of common used triple therapy for Helicobacter pylori infection (less than 80%).

Objective: To determine the optimal pre-concommitant treatment length for rabeprazole based sequential-concomitant hybrid therapies for adults infected with Helicobacter pylori in Eastern Taiwan.

Design: Randomized, open-label, prospective controlled trial.

Patients: 231 patients with dyspepsia or peptic ulcers and infected by Helicobacter pylori.

Measurements: 13C-urea breath test, upper endoscopy, histologic evaluation, rapid urease test, bacterial culture, assessment of antibiotic resistance and CYP2C19 genotype of host.

Intervention: 231 patients with Helicobacter pylori infection are recruited and randomly assigned to receive one of the following therapeutic schemes: group 1, 14-days hybrid therapy: rabeprazole 20mg bid + amoxicillin 1g bid treated for 7 days, then rabeprazole 20mg bid + amoxicillin 1g bid + clarithromycin 0.5g bid + metronidazole 0.5g bid for other 7 days; group 2, 12-days hybrid therapy: rabeprazole 20mg bid + amoxicillin 1g bid treated for 5 days, then rabeprazole 20mg bid + amoxicillin 1g bid + clarithromycin 0.5g bid + metronidazole 0.5g bid for other 7 days; group 3, 10-days hybrid therapy: rabeprazole 20mg bid + amoxicillin 1g bid treated for 3 days, then rabeprazole 20mg bid + amoxicillin 1g bid + clarithromycin 0.5g bid + metronidazole 0.5g bid for other 7 days. Repeat upper endoscopy for histologic evaluation, rapid urease test or 13C-urea breath test after 4 week of treatment to assess the treatment result. The influence on the hybrid therapies of antibiotic resistance of Helicobacter pylori and CYP2C19 genotype of host were determined.

Expected results: The rabeprazole based sequential-concomitant therapies for eradication of Helicobacter pylori is very effective, and the outcome is not affected by antibiotic resistance of Helicobacter pylori and CYP2C19 genotype of host.

ELIGIBILITY:
Inclusion Criteria:

* Patient proved with infection of H. pylori in gastric mucosa (at least two of four tests positive)

Exclusion Criteria:

* woman in breast feeding or pregnancy.
* allergy to drugs used in study.
* previously treated for H. pylori.
* intolerance to fructose, lactose.
* patients with hematologic, brain or spinal disorders
* patients under 20 years old
* patients under aspirin or clopidogrel
* patients with history of gastric cancer or gastric resection operation.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 4 weeks after complete use of drug for treatment
  A negative post-treatment 13C-urea breath test result at more than 4 weeks after complete use of drug for treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Cheh CHEN, MD, Principal Investigator — Buddhist Tzu Chi General Hospital
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan, Taiwan